CLINICAL TRIAL: NCT03770962
Title: One Plus One Equals Two - Will That do? A Randomized Controlled Trial to Evaluate Collegial Midwifery Practice to Prevent Perineal Trauma
Brief Title: One Plus One Equals Two, Will That do?
Acronym: Oneplus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/476
Record Dates: First submitted 2018-11-28; First posted 2018-12-10 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Sphincter (Anal); Perineal Rupture, Obstetric; Perineal Tear; Pelvic Floor Disorders; Experience, Life; Second Stage of Labor
Keywords: Midwifery intervention; Birth experience; Obstetric anal sphincter injuries; Perineal tears
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The statistician who performs the statistical analysis will be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two midwives (Experimental): Two midwives will be present during the active phase of the second stage and the birth of the baby. "Midwife no 1" is the midwife who has been responsible for the care of the woman and "midwife no 2" will observe the birth or give any assistance needed.
  Interventions: Behavioral: Two midwives
- One midwife (No Intervention): This is standard care. One midwife is responsible for the care of the woman and her unborn baby during labor and birth.

INTERVENTIONS:
Behavioral: Two midwives — Two midwives will be present during the active phase of the second stage and the birth of the baby. "Midwife no 1" is the midwife who has been responsible for the care of the woman and "midwife no 2" will assist her.
  Arms: Two midwives

SUMMARY:
A new clinical practice to reduce perineal trauma has been adopted by many maternity wards in Sweden. This practice involves collegial midwifery assistance during the second stage of labor and the birth of the baby. The midwife responsible for the birth is the primary carer of the woman and the second midwife observes the birth or assists the primary midwife if asked to. The hypothesis is that the presence and support of an extra midwife will reduce severe perineal trauma (trauma to the anal sphincter (OASI)).

The objective of this trial is to evaluate whether collegial midwifery assistance during the second stage reduces perineal trauma grade III-IV.

DETAILED DESCRIPTION:
Most women sustain some form of perineal trauma when giving birth vaginally. Perineal injuries are classified as grade I-IV. A first-degree tear only includes perineal skin or mucosa, whereas a second-degree tear includes muscles in the perineal body. A tear involving a part or the whole of the anal sphincter muscle complex is graded III-IV. Data from the Swedish National Birth Register show that 4% of first-time mothers suffered a tear affecting the anal sphincter. National registers in Sweden only collect data on severe perineal trauma affecting the anal sphincter but in a recent regional Swedish study 78% of the primiparous women experienced second-degree tears. The consequences of second-degree tears and severe perineal trauma are pain, dyspareunia, and an increased risk of symptomatic pelvic organ prolapse later in life. A severe consequence of perineal trauma is anal incontinence, mainly caused by tears affecting the anal sphincter muscle. However, second-degree tears may also lead to anal incontinence. This may be related to a lack of support from the perineal body due to poor repair. Furthermore, perineal trauma is known to be misclassified, with consequent under-reporting of injuries affecting the anal sphincter complex.

Risk factors for severe perineal trauma (grade III-IV) are giving birth vaginally for the first time, having an assisted vaginal birth, giving birth vaginally after a previous caesarean section, or giving birth to a baby that weighs more than 4000 g, and the risk increases with age. Some of the midwifery care methods used to prevent perineal injuries have been evaluated in clinical trials but there are still gaps in the investigator's knowledge. Even if scientific evidence is lacking for most of the preventive strategies used by midwives except for warm compresses held at the perineum, midwives believe that a slow and controlled birth is a key factor in prevention. Several studies indicate that a combination of strategies can be effective in preventing perineal trauma. Giving birth is a profound experience for the woman and her partner and an experience that has significance for the woman all her life. The second stage is considered to be the most stressful part of the labor for the woman and her unborn baby, and consequently also for the midwife. Despite this, there is still a lack of knowledge about how women experience the second stage and the methods midwives use to facilitate birth and prevent perineal trauma. Traditionally midwives have asked colleagues for a second opinion or to assist in complicated situations, or in obstetric emergencies. Recently a new clinical practice has been introduced in approximately 50% of the maternity wards in Sweden to reduce severe perineal trauma. This procedure involves two midwives attending the woman during the second stage of labor. The midwife responsible for the birth calls for the second midwife when the active phase of the second stage has started and the presenting part of the baby is visible. The second midwife observes the birth and can assist the midwife responsible for the birth if needed. An unpublished survey from one maternity ward in Sweden showed that most of the midwives appreciated this way of working but were uncertain as to whether it actually reduced the prevalence of severe perineal trauma. Furthermore, this clinical practice might have negative side-effects or unintended consequences. The maternity wards that practise this method have not increased the number of midwives. It could be argued that there is a risk that other women in labor will be left unattended for longer periods when two midwives assist at births. How midwives share the responsibility and communicate are factors that needs to be evaluated scientifically.

The objective of this trial is to evaluate whether collegial midwifery assistance during the second stage reduces perineal trauma grade III-IV.

Data from the National Birth Register show that 4.1% of first-time mothers suffered severe perineal trauma (OASI) in Sweden 2017. To be able to detect a reduction from 4.1 to 2.0% (50% reduction) with 80% power and a 95% level of significance, 1052 women in each group will be needed. The 50% reduction is based on regional figures after a change in practice and is therefore clinically significant. Allowing for a possible 40% drop-out rate including possible cases of obstetric emergencies where another midwife will be needed regardless of randomization, this will result in 2946 women in total. To ensure that there are no adverse side-effects of the intervention interim analyses will be performed every 6 months until the end of the trial. In the interim analysis, the distribution of the intervention and standard care will be estimated among women with no perineal tears, women diagnosed with a third- or fourth-degree tear (OASI), and neonatal outcome (apgar score at 5 minutes and arterial blood gas from the nuchal cord).

Women will be asked to participate in the trial when arriving to the maternity ward. The randomization will take place when the woman enters the second stage. It will not be possible to blind either women or midwives in this study. The participants will be randomly allocated (1:1) to the intervention group or to the standard care group. To allow for equal distribution between the groups, block randomization in blocks of ten (five to the intervention and five to the control group) will be used.

After the birth the tear will be diagnosed together with a midwife or an obstetrician who has not been involved in the birth. Tears will be sutured according to the guidelines at each participating study site. The midwife responsible for the birth will complete a questionnaire which will contain questions regarding the woman; labor and birth variables, methods of preventing perineal trauma, questions regarding the baby, diagnosis of the tear and how the tear was sutured. If a second midwife has been present during the second stage (intervention) the responsible midwife will also complete questions on the assistance she got from the second midwife and how this assistance was experienced. Data will also be retrieved from the participating women's records by using the local database of each study site. When the intervention has taken place the second midwife will also complete a questionnaire.

The women in the trial will be sent a questionnaire one month and one year after the birth. The follow-up questionnaire after one month will contain questions regarding their experience of the intervention and their experience of the methods used during the second stage and women's well-being (EPDS, Pain relief, sexual intercourse resumption, breastfeeding initiation), after birth.

For the one-year follow-up the following validated questionnaires will be used: Pelvic Floor Impact Questionnaire (PFIQ7), Pelvic Floor Distress Inventory - short form (PFDI-20), Pelvic Organ Prolapse/Urinary Incontinence Sexual Function Questionnaire (PISQ-12) Female Sexual Function Index FSFI, Edinburgh Postnatal Depression Scale (EPDS) and breastfeeding duration.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women
* Primiparous women with one previous cesarean section who plan for a vaginal birth
* >37+0 week of gestational age

Exclusion Criteria:

* Multiparous women
* Twin pregnancies
* Planned breech delivery
* Preterm birth
* Nulliparous women with planned elective cesarean section
* Not able to understand oral and written information regarding the study

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3058 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Number of women with obstetric anal sphincter injury | 4 hour
  Tear of the external and/or internal anal sphincter at any degree, ICD-10 O70.2 and O70.3.

SECONDARY OUTCOMES:
Number of women with perineal tear grade II | 4 hour
  Tear of the muscles of the perineum and/or deeper vaginal tears. ICD-10 O70.1
Number of women with postpartum bleeding | 6 hour
  Postpartum bleeding in millilitres evaluated 6 hours after birth. ICD-10 O72.0, O72.1 (O72.1a, O72.1b)
Birthposition at the time of birth | 2 hours
  The position of the woman when giving birth as recorded in the local birth register
Number of women with an episiotomy | 4 hour
  Number of women who had an episiotomy performed during birth
Number of women with perineal injury subtypes | 4 hour
  Labial lacerations, periurethral tears, perinal tears grade I, and superficial vaginal tears. ICD-10 070.0
Apgar scores at birth, 1 and 5 min after birth | 10 minutes
  Apgar score assessed by the midwife a 1,5.10 minutes after the baby is born
pH in umbilical artery | Blood sample is drawn from the umbilical cord within 1 minute after the birth of the baby and evaluated within 30 minutes
  Arterial pH in the umbilical cord
Breastfeeding within 2 hours after birth | 2 hours
  Number of women who breastfeed within 2 hours after birth
Number of women with an assisted Instrumental delivery | Recorded after birth (2 hours)
  Number of women with an instrumental delivery (vacuum extraction or forceps)
Midwives experiences of the intervention | One month
  Midwives no 1 and no 2 will complete a study record after birth. The study record will contain question regarding what midwife no 2 assisted with during the second stage of labour and how it was perceived by midwife no 1
Women's experiences of midwifery methods used during the second stage of labor | One month
  Study specific questions sent to women one month after the birth. A questionnaire with questions regarding midwifery methods used (YES or NO) during the second stage of labor and how they were perceived by the participating women. Questions with Likert scale answers.
Number of women with urinary incontinence 1 year after birth | 1 year
  Questionnaire 12 months after the birth. Pelvic Floor Impact Questionnaire (PFIQ) will be used.
Number of women with anal incontinence 1 year after birth | 1 year
  Questionnaire 12 months after the birth. Pelvic Floor Impact Questionnaire (PFIQ) will be used
Female Sexual Function Index (FSFI) one year after birth | 1 year
  Questionnaire 12 months after the birth. Sexual Function Questionnaire (FSFI) will be used
Number of women with pelvic organ prolapse symptoms 1 year after birth | 1 year
  Questionnaire 12 months after the birth. Pelvic Floor Impact Questionnaire (PFDI-20) will be used
Number of women who scored 12 point or above on the Edinburgh Postnatal Depression Scale | one month
  Depressive symptoms 1 month after birth as reported on the Edinburgh Postnatal Depression Scale (EPDS)
Number of women who scored 12 point or above on the Edinburgh Postnatal Depression Scale | 1 year
  Depressive symptoms 1 year after birth as reported on the Edinburgh Postnatal Depression Scale (EPDS)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Rubertsson, Professor, Principal Investigator — Institution of Health Sciences, The Faculty of Medicine, Lund University; Pia Teleman, Ass.prof, Study Chair — Region Skåne SUS
Locations (4):
- Sweden (4):
  - Lund Delivery Ward, SUS Region Skåne, Lund, Skåne County
  - Malmö Delivery Ward, SUS Region Skåne, Malmo, Skåne County
  - Karlstad delivery ward, Karlstad, Värmland County
  - PO Pregnancy and Birth, Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baghestan E, Irgens LM, Bordahl PE, Rasmussen S. Trends in risk factors for obstetric anal sphincter injuries in Norway. Obstet Gynecol. 2010 Jul;116(1):25-34. doi: 10.1097/AOG.0b013e3181e2f50b. PMID 20567164
- [Background] Edqvist M, Hildingsson I, Mollberg M, Lundgren I, Lindgren H. Midwives' Management during the Second Stage of Labor in Relation to Second-Degree Tears-An Experimental Study. Birth. 2017 Mar;44(1):86-94. doi: 10.1111/birt.12267. Epub 2016 Nov 14. PMID 27859542
- [Background] Macarthur AJ, Macarthur C. Incidence, severity, and determinants of perineal pain after vaginal delivery: a prospective cohort study. Am J Obstet Gynecol. 2004 Oct;191(4):1199-204. doi: 10.1016/j.ajog.2004.02.064. PMID 15507941
- [Background] Rathfisch G, Dikencik BK, Kizilkaya Beji N, Comert N, Tekirdag AI, Kadioglu A. Effects of perineal trauma on postpartum sexual function. J Adv Nurs. 2010 Dec;66(12):2640-9. doi: 10.1111/j.1365-2648.2010.05428.x. Epub 2010 Aug 23. PMID 20735499
- [Background] Tegerstedt G, Miedel A, Maehle-Schmidt M, Nyren O, Hammarstrom M. Obstetric risk factors for symptomatic prolapse: a population-based approach. Am J Obstet Gynecol. 2006 Jan;194(1):75-81. doi: 10.1016/j.ajog.2005.06.086. PMID 16389012
- [Background] Woodman PJ, Graney DO. Anatomy and physiology of the female perineal body with relevance to obstetrical injury and repair. Clin Anat. 2002 Aug;15(5):321-34. doi: 10.1002/ca.10034. PMID 12203375
- [Background] Schei B, Johannessen HH, Rydning A, Sultan A, Morkved S. Anal incontinence after vaginal delivery or cesarean section. Acta Obstet Gynecol Scand. 2019 Jan;98(1):51-60. doi: 10.1111/aogs.13463. Epub 2018 Oct 29. PMID 30204238
- [Background] Andrews V, Sultan AH, Thakar R, Jones PW. Occult anal sphincter injuries--myth or reality? BJOG. 2006 Feb;113(2):195-200. doi: 10.1111/j.1471-0528.2006.00799.x. PMID 16411998
- [Background] Raisanen S, Vehvilainen-Julkunen K, Cartwright R, Gissler M, Heinonen S. A prior cesarean section and incidence of obstetric anal sphincter injury. Int Urogynecol J. 2013 Aug;24(8):1331-9. doi: 10.1007/s00192-012-2006-6. Epub 2012 Dec 5. PMID 23212242
- [Background] Raisanen SH, Vehvilainen-Julkunen K, Gissler M, Heinonen S. Lateral episiotomy protects primiparous but not multiparous women from obstetric anal sphincter rupture. Acta Obstet Gynecol Scand. 2009;88(12):1365-72. doi: 10.3109/00016340903295626. PMID 19852569
- [Background] Elvander C, Ahlberg M, Edqvist M, Stephansson O. Severe perineal trauma among women undergoing vaginal birth after cesarean delivery: A population-based cohort study. Birth. 2019 Jun;46(2):379-386. doi: 10.1111/birt.12402. Epub 2018 Oct 22. PMID 30350424
- [Background] Aasheim V, Nilsen ABV, Reinar LM, Lukasse M. Perineal techniques during the second stage of labour for reducing perineal trauma. Cochrane Database Syst Rev. 2017 Jun 13;6(6):CD006672. doi: 10.1002/14651858.CD006672.pub3. PMID 28608597
- [Background] Laine K, Pirhonen T, Rolland R, Pirhonen J. Decreasing the incidence of anal sphincter tears during delivery. Obstet Gynecol. 2008 May;111(5):1053-7. doi: 10.1097/AOG.0b013e31816c4402. PMID 18448735
- [Background] Basu M, Smith D, Edwards R; STOMP project team. Can the incidence of obstetric anal sphincter injury be reduced? The STOMP experience. Eur J Obstet Gynecol Reprod Biol. 2016 Jul;202:55-9. doi: 10.1016/j.ejogrb.2016.04.033. Epub 2016 Apr 30. PMID 27164486
- [Background] Basu M, Smith D. Long-term outcomes of the Stop Traumatic OASI Morbidity Project (STOMP). Int J Gynaecol Obstet. 2018 Sep;142(3):295-299. doi: 10.1002/ijgo.12565. Epub 2018 Jul 5. PMID 29885253
- [Background] Simkin P. Just another day in a woman's life? Women's long-term perceptions of their first birth experience. Part I. Birth. 1991 Dec;18(4):203-10. doi: 10.1111/j.1523-536x.1991.tb00103.x. PMID 1764149
- [Background] Kopas ML. A review of evidence-based practices for management of the second stage of labor. J Midwifery Womens Health. 2014 May-Jun;59(3):264-76. doi: 10.1111/jmwh.12199. PMID 24850283
- [Derived] Edqvist M, Ajne G, Teleman P, Tegerstedt G, Rubertsson C. Postpartum perineal pain and its association with sub-classified second-degree tears and perineal trauma-A follow-up of a randomized controlled trial. Acta Obstet Gynecol Scand. 2024 Nov;103(11):2314-2323. doi: 10.1111/aogs.14938. Epub 2024 Aug 16. PMID 39150169
- [Derived] Haggsgard C, Edqvist M, Teleman P, Tern H, Rubertsson C. Impact of collegial midwifery assistance during second stage of labour on women's experience: a follow-up from the Swedish Oneplus randomised controlled trial. BMJ Open. 2024 Jul 27;14(7):e077458. doi: 10.1136/bmjopen-2023-077458. PMID 39067883
- [Derived] Haggsgard C, Rubertsson C, Teleman P, Edqvist M. Informed consent to midwifery practices and interventions during the second stage of labor-An observational study within the Oneplus trial. PLoS One. 2024 Jun 12;19(6):e0304418. doi: 10.1371/journal.pone.0304418. eCollection 2024. PMID 38865296
- [Derived] Edqvist M, Dahlen HG, Haggsgard C, Tern H, Angeby K, Tegerstedt G, Teleman P, Ajne G, Rubertsson C. One Plus One Equals Two-will that do? A trial protocol for a Swedish multicentre randomised controlled trial to evaluate a clinical practice to reduce severe perineal trauma 1. Trials. 2020 Nov 23;21(1):945. doi: 10.1186/s13063-020-04837-7. PMID 33225972
- See also: The Swedish birthregister. Annual Report 2017 (Swedish) — https://www.medscinet.com/GR/uploads/hemsida/dokumentarkiv/GR_%C3%85rsrrapport_2017_4.0.pdf
- See also: Midwives' experiences of collegial presence during the second stage of labour (Swedish) — http://www.diva-portal.org/smash/get/diva2:901989/FULLTEXT01.pdf
- See also: The Management of Third- and Fourth-Degree Perineal Tears. RCOG Green-top Guideline No.29 — https://www.rcog.org.uk/globalassets/documents/guidelines/gtg-29.pdf

DOCUMENTS (1):
  • Study Protocol (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT03770962/Prot_001.pdf